CLINICAL TRIAL: NCT03963635
Title: Novel Diagnostics for Early Lyme Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: MicroB-plex, Inc. (Industry)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: 12251305
Record Dates: First submitted 2019-05-23; First posted 2019-05-28 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Lyme Disease
Keywords: Lyme Disease; Borrelia burgdorferi; Antibody Secreting Cells; Diagnostics; Early Diagnosis; Treatment Outcome; Health Volunteers; Adult
MeSH Terms: conditions — Lyme Disease; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Anti-coagulated whole blood, Serum, Peripheral Blood Mononuclear Cells
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lyme Infected: Subjects presenting with suspected Lyme Disease
  Interventions: Diagnostic Test: MicroB-plex Lyme Immunoassay
- Controls: Subjects with no known Lyme Disease, past or present
  Interventions: Diagnostic Test: MicroB-plex Lyme Immunoassay

INTERVENTIONS:
Diagnostic Test: MicroB-plex Lyme Immunoassay — Subject's blood and clinical data are collected to develop a diagnostic immunoassay

SUMMARY:
There are more than 300,000 new cases of Lyme disease every year in the US. Lyme disease is a dangerous bacterial infection transmitted by tick bites and it becomes increasingly severe as the infection progresses. Definitive diagnosis is based on serum-based tests that have fundamental limitations: 1) current tests cannot detect early infections so patients do not receive antibiotic therapy until the infection has progressed, and 2) there is no way to measure if antibiotic therapy has been successful. MicroB-plex will address these two unmet clinical needs by introducing a novel, blood-based diagnostic method that will enable clinicians to diagnose infections earlier and to monitor the success of their interventions.

DETAILED DESCRIPTION:
Lyme disease is the most commonly reported arthropod-borne infection in the US with recent CDC estimates eclipsing 300,000 new cases in 2013. In addition to growing in frequency, the infections have a complex and increasingly severe course. Beginning with mild flu-like symptoms and frequently a signature bull's-eye rash, erythema migrans, Lyme disease can progress to severe articular, neurological and cardiac symptoms, most of which are preventable with early antibiotic therapy. Leading investigators have identified two major shortcomings to the current serology-based methods for the definitive diagnosis of Early Localized Lyme disease. First, the clinical sensitivity in the first four weeks is poor, under 50% at the time of symptom onset, so many patients remain undiagnosed or unconfirmed until the disease has had time to progress. Second, serum antibody levels remain elevated long after the infection has been resolved making the monitoring of therapeutic success or diagnosis of re-infection virtually impossible. MicroB-plex will address these shortcomings by using a novel sample matrix from circulating antibody secreting cells (ASC) for diagnosis of Lyme disease. This novel matrix is MENSA (medium enriched for newly synthesized antibody). In this study, MicroB-plex and its clinical collaborators will test whether MENSA is effective in early Lyme diagnostic (within the first 2 weeks) and if this new approach will track therapeutic success.

ELIGIBILITY:
Inclusion Criteria:

1. Human adults at least 21 years of age and no more than 80 years of age at the time of screening.
2. Have the ability to understand the requirements of the study, provide written informed consent (including consent for the use and disclosure of research-related health information), and comply with the study protocol procedures (including required study visits).
3. High clinical suspicion of acute Lyme disease, with symptoms seven days or less.
4. Must have erythema migrans rash and physician diagnosis of early Lyme disease.
5. Brief history and physical exam will be obtained during the study visit.
6. Be willing to return to our clinic for up to nine visits and blood draws over a one-year period.
7. People who do not have Lyme disease, but want to participate as healthy controls (one time visit)

Exclusion Criteria:

1. Have poor venous access.
2. Have received any immunosuppressive therapy including biologics or recent course of steroids, or recent chemotherapy.

   1. Anti-TNF therapy (eg, adalimumab, etanercept, infliximab).
   2. Intravenous (IV) cyclophosphamide
   3. Interleukin-1 receptor antagonist (anakinra).
   4. Intravenous immunoglobulin (IVIG).
   5. High dose prednisone or equivalent (> 100 mg/day).
   6. Plasmapheresis.
   7. Any new immunosuppressive/immunomodulatory agent
   8. Any steroid injection (eg, intramuscular, intraarticular, or intravenous).
3. On treatment for Lyme disease greater than seven days
4. Recent chemotherapy
5. History of solid organ transplant
6. History of autoimmune disorders (SLE, Rheumatoid arthritis, Scleroderma, etc.)
7. History of inflammatory muscle disease (polymyositis, dermatomyositis, etc.)
8. History of inflammatory bowel disease (Crohn's disease, Ulcerative colitis, etc.)
9. History of HIV infection
10. Received a Lyme disease vaccine in the past
11. History of prior Lyme disease infection in the past
12. Have any condition that, in the opinion of the principal investigator, would significantly increase the risk for the subject.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult humans with a strong clinical suspicion of acute Lyme disease, with symptoms seven days or less. Subjects will be recruited from medical centers residing in Maryland.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of EM positive patients who become MicroB-plex Lyme test positive prior to seroconversion | Within 14 days of enrollment
  MicroB-plex Lyme Test, that measures anti-Lyme antibodies in MENSA, becomes positive prior to conventional Lyme immunoassays that measure antibodies in serum, resulting in earlier diagnosis
Percentage of treated EM positive patients who become MicroB-plex Lyme test negative prior to their decline in serum | Up to one year from enrollment
  MicroB-plex Lyme Test, that measures anti-Lyme antibodies in MENSA, becomes negative with successful treatment, prior to a decline in serum antibody level in conventional immunoassays, providing an earlier measure of effective therapy

SECONDARY OUTCOMES:
Percentage of treated EM positive patients who remain MicroB-plex Lyme test positive following treatment | Up to one year from enrollment
  MicroB-plex Lyme Test, that measures anti-Lyme antibodies in MENSA, remains positive with treatment failure

CONTACTS AND LOCATIONS:
Overall Officials: John L Daiss, PhD, Principal Investigator — MicroB-plex, Inc.; Frances E Lee, MD, Principal Investigator — MicroB-plex, Inc.
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No